CLINICAL TRIAL: NCT04035616
Title: Evaluation of the Efficacy of Probiotics in Treating Constipation in Elderly Patients With Multiple Chronic Co-morbidities: a Randomized Control Trial
Brief Title: Probiotics in Elderly Patients With Medical Conditions
Acronym: Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2016-417); NMRR-19-1761-49477 (Registry Identifier: The National Medical Registry of Malaysia)
Record Dates: First submitted 2019-07-17; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Aging; Constipation; Multi-Core Disease
Keywords: microbial cell preparation; Hexbio®; probiotics; elderly; chronic medical conditions; constipation,
MeSH Terms: conditions — Constipation; Minicore Myopathy with External Ophthalmoplegia

STUDY DESIGN:
Intervention Model Description: The subjects received either the probiotics or a placebo.
Who Masked: Participant, Investigator
Masking Description: Both investigators and patients were unaware of the assignment and were blinded to the labelling process performed by the sample supplier. The patients were randomly allocated to one of two groups; those who received sample labelled A or B. Emergency code break were kept at the manufacturing factory and no code break was needed throughout the trial duration. Both the MCP and placebo were manufactured and supplied by B-Crobes Laboratory Sdn. Bhd. as powder in identical sachets and labelled as A and B. Investigators have no contact with the manufacturing staffs at any point during the trial process. Following data analysis, unblinding was performed to complete the study process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo were manufactured and supplied by B-Crobes Laboratory Sdn. Bhd. as powder in identical sachets with active comparator and labelled as A
  Interventions: Other: placebo
- Hexbio® MCP (Active Comparator): The treatment sample is labelled as B.This is an orange-flavoured, granulated microbial cell preparation containing 30 billion colony forming units (cfu) of Lactobacilli and Bifidobacteria strains: Lactobacillus acidophilus BCMC® 12130, Lactobacillus casei BCMC® 12313, Lactobacillus lactis BCMC® 12451, Bifidobacterium bifidum BCMC® 02290, Bifidobacterium infantis BCMC®02129, Bifidobacterium longum BCMC® 02120. The placebo sample was similar in appearance and taste, but contained no microbial cells.
  Interventions: Dietary Supplement: microbial cell preparation [MCP]

INTERVENTIONS:
Dietary Supplement: microbial cell preparation [MCP] — active microbial cell preparation
  Other Names: Hexbio®
  Arms: Hexbio® MCP
Other: placebo — inactive ingredient
  Arms: Placebo

SUMMARY:
Study of efficacy of probiotic in older patients with multiple co-morbidites and constipation

DETAILED DESCRIPTION:
Background and aims:

Probiotics are known to have a beneficial effect on the management of constipation. Thus, the current study objective was to evaluate the impact of a microbial cell preparation (MCP) (Hexbio®; comprising Bifidobacterium and Lactobacillus strains) on stool frequency, consistency, and constipation-related symptoms in elderly patients with multiple chronic medical conditions.

ELIGIBILITY:
Inclusion Criteria:

-clinical diagnosis of constipation

Exclusion Criteria:

* Parkinson's disease,
* spinal cord lesions
* post radiation strictures
* on calcium supplements of greater than 1,500 mg per day
* immune-deficiency
* critical illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
changes in stool output frequency | 7 days
  numerical scale 0-100 used, 0= nil (worst), 100= good, medium score was used for data interpratation
changes in stool consistency | 7 days
  The Bristol Stool scale was used, scale type 1 to 7, type 1 = hard stool and type 7=entirely liquid stool, medium score was used for data intepretation

SECONDARY OUTCOMES:
patients' perceptions of an improvement in their constipation-related symptoms 1 | 7 days
  straining: likert score of 0 to 10 was used, 0=no straining, 10= worst straining
patients' perceptions of an improvement in their constipation-related symptoms 2 | 7 days
  sensation of incomplete evacuation: likert score of 0 to 10 was used, 0= total incomplete evacuation, 10=complete evacuation
patients' perceptions of an improvement in their constipation-related symptoms 3 | 7 days
  sensation of ano-rectal obstruction/blockage: likert score of 0 to 10 was used, 0=complete obstruction, 10= complete relieved
patients' perceptions of an improvement in their constipation-related symptoms 4 | 7 days
  Need of manual evacuation to aid defeacation: likert score of 0 to 10 was used, 0=no evacuation needed, 10=total evacuation needed

CONTACTS AND LOCATIONS:
Overall Officials: hayati Yaakup, MBBS, Principal Investigator — National University of Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia Medical Faculty, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghafar MYA, Yaakup H, Ali RAR, Shah SA. Evaluation of the Efficacy of Probiotics (MCP(R) BCMC(R) Strains) Treating Constipation in Elderly Patients with Multiple Chronic Co-Morbidities: A Randomized Control Trial. J Nutr Health Aging. 2020;24(10):1066-1072. doi: 10.1007/s12603-020-1494-1. PMID 33244562

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04035616/Prot_SAP_000.pdf